CLINICAL TRIAL: NCT04597333
Title: Comparison of Cervical Ripening Balloon Versus 2nd Dinoprostone Insert for Labor Induction in Women With a Failed 1st Attempt of Induction With Dinoprostone.
Brief Title: Labor Induction After Failed Induction With Dinoprostone.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0009-20-RMB
Record Dates: First submitted 2020-10-15; First posted 2020-10-22 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Induction of Labor Affected Fetus / Newborn
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2nd Dinoprostone. (Active Comparator): Women induced with a second dinoprostone insert.
  Interventions: Drug: Dinoprostone
- Cervical ripening balloon. (Active Comparator): Women induced with a cervical ripening balloon.
  Interventions: Device: Cervical ripening balloon.

INTERVENTIONS:
Drug: Dinoprostone — Dinoprostone vaginal insert.
  Arms: 2nd Dinoprostone.
Device: Cervical ripening balloon. — Double lumen cervical ripening balloon.
  Arms: Cervical ripening balloon.

SUMMARY:
Women after induction of labor with a dinoprostone insert will be evaluated after 24 hours from the beginning of labor induction. Women with a BISHOP score of less than 5 will be randomized to 1 of 2 groups. Induction with a cervical ripening balloon versus induction with a 2nd dinoprostone insert.

DETAILED DESCRIPTION:
Nulliparous women with obstetric indications for induction of labor who were induced with a dinoprostone insert and failed to go into labor after 24 hours from the beginning of labor induction and a BISHOP score of less than 5 will receive a thorough explanation regarding the study and sign informed consent. The eligible women will be randomized to 1 of 2 groups. Induction with a cervical ripening balloon versus induction with a 2nd dinoprostone insert. Relevant demographic and medical information will be gathered from the patients' electronic files.

ELIGIBILITY:
Inclusion Criteria:

* Women after induction of labor with Dinoprostone.
* BISHOP score of under 5 after 1st induction attempt.
* Nulliparous women.

Exclusion Criteria:

* Women after induction of labor with a cervical ripening balloon.
* BISHOP score of over 5 after 1st induction attempt.
* Multiparous women.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female.
Enrollment: 144 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Delivery within 24 hours. | From the time of induction up to 24 hours from induction.
  Rate of delivery in 24 hours.
Time to delivery. | From the time of induction up to 120 hours from induction.
  The number of hours it takes to deliver.

SECONDARY OUTCOMES:
Mode of delivery. | From the time of induction up to 120 hours from induction.
  Vaginal and cesarean delivery rates.
Uterine revision. | From the time of induction up to 120 hours from induction.
  The rate of uterine revision postpartum.
Postpartum hemorrhage. | From the time of induction up to 120 hours from induction.
  The rate of postpartum hemorrhage.
Chorioamnionitis. | From the time of induction up to 120 hours from induction.
  The rate of chorioamnionitis.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam health care campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No